CLINICAL TRIAL: NCT03608852
Title: Bad is Stronger Than Good: Unconventional Financial Incentives for Smoking Cessation
Brief Title: Unconventional Financial Incentives for Smoking Cessation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gregory Holt, Internal Medicine, Miami VA Healthcare System
Other Study IDs: 1160736-1
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Banked-money group: This group will have $50 placed in a 'bank account' for every clinic visit where their tests reveal abstinence from smoking. As a modified commitment contract, the Banked-Money Group can only withdraw the accrued money at the end of the trial if they complete the trial by quitting smoking for the entire 6 months.
- Reward group: This group will directly receive $50 for every clinic visit where their tests reveal abstinence from smoking.

SUMMARY:
The proposed study is a randomized study of actively smoking veterans cared for at the Miami VA Medical Center. Subjects are randomized into 2 groups and will all receive a regimen of nicotine replacement therapy (NRT) standardized to their smoking habit. Subjects are followed biweekly for smoking cessation by using biochemical tests (exCO and COHb) to determine smoking abstinence. The first group called the Banked-Money Group will have $50 placed in a 'bank account' for every clinic visit where their tests reveal abstinence from smoking. As a modified commitment contract, the Banked-Money Group can only withdraw the accrued money at the end of the trial if they complete the trial by quitting smoking for the entire 6 months. The second group called the Reward Group will directly receive $50 for every clinic visit where their tests reveal abstinence from smoking.

ELIGIBILITY:
Inclusion Criteria:

Enrollment criteria include subjects 18 years of age or older, currently smoking at least a half a pack of cigarettes a day, who have at least a ten-pack year smoking history, are interested in quitting smoking, agree to submit to exhaled breath and ABG analysis and have reliable means of visiting the clinic every two weeks. Subjects must be able to tolerate NRT including patches and lozenges and meet with the VA smoking cessation counselor.

Exclusion Criteria:

Subjects will not be enrolled if they are currently taking varenicline as the VA disallows concurrent use of varenicline and NRT.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The goal of this study is to enroll 36 active smokers
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation rate | 1 year
  The primary outcome for this study is to compare smoking cessation rates between smokers who received one of two financial incentive strategies in addition to standard of care NRT and counseling.

SECONDARY OUTCOMES:
Household income | 1 year
  We will determine whether household income affect quit rates.
Smoking habits | 1 year
  We will determine whether smoking habits affect quit rates.
Nicotine dependence | 1 year
  We will determine whether nicotine dependence affect quit rates.
Nicotine withdrawal symptoms | 1 year
  We will determine whether nicotine withdrawal symptoms affect quit rates.
Anxiety / Depression | 1 year
  We will determine whether anxiety and / or depression affect quit rates.

IPD SHARING:
Plan to Share IPD: No